CLINICAL TRIAL: NCT03597698
Title: Ill-health Related Jobloss
Brief Title: Ill-health Related Job Loss
Acronym: jobloss
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Université Montpellier (Other); Occupational Health Center, Montpellier, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0021
Record Dates: First submitted 2018-02-22; First posted 2018-07-24 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-02

CONDITIONS: Job Loss Noticed by the Occupational Physicians
Keywords: job loss; unfit for a job

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The current study aimed to estimate the one-year incidence of unfitness for the job in an occupational health service, and to describe their aetiology and the characteristics of the unfit employees

ELIGIBILITY:
Inclusion Criteria:

- to be followed-up in the occupational health center

Exclusion criteria:

- civil servants

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all the workers followed up in an occupational health center of Montpellier
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2014-12-01 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
number of job loss | 1 day
  number of job loss related to poor health

SECONDARY OUTCOMES:
highlight trades or sectors associated with increased risk of medical incapacity | 1 day
  identify occupations or sectors associated with an increased risk of medical incapacity, regardless of the socio-demographic characteristics (including age and sex) of employees in the occupation

CONTACTS AND LOCATIONS:
Overall Officials: Francois Xavier LESAGE, MD, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC